CLINICAL TRIAL: NCT00655369
Title: PD 0200390 Dose-Ranging Trial: A Randomized, Double-Blind, Parallel Group, Placebo-Controlled, Multicenter Outpatient Trial of PD 0200390 in Adults With Nonrestorative Sleep
Brief Title: A Double-blind, Parallel Group, Placebo-Controlled Outpatient Trial of PD 00200390 in Adults With Nonrestorative Sleep
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: A4251033
Record Dates: First submitted 2008-04-03; First posted 2008-04-09 (Estimated); Last update posted 2012-07-25 (Estimated); Status verified 2012-07

CONDITIONS: Nonrestorative Sleep
MeSH Terms: interventions — (1-aminomethyl-3,4-dimethylcyclopentyl)acetic acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- 15 mg (Experimental)
  Interventions: Drug: PD 0200390
- 25 mg (Experimental)
  Interventions: Drug: PD 0200390
- 35 mg (Experimental)
  Interventions: Drug: PD 0200390
- 5 mg (Experimental)
  Interventions: Drug: PD 0200390
- 50 mg (Experimental)
  Interventions: Drug: PD 0200390
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PD 0200390 — oral 15 mg daily dose, 3 capsules per dose during a six week treatment period.
  Arms: 15 mg
Drug: PD 0200390 — oral 25 mg daily dose, 3 capsules per dose during a six week treatment period.
  Arms: 25 mg
Drug: PD 0200390 — oral 35 mg daily dose, 3 capsules per dose during a six week treatment period.
  Arms: 35 mg
Drug: PD 0200390 — oral 5 mg daily dose, 3 capsules per dose during a six week treatment period.
  Arms: 5 mg
Drug: PD 0200390 — oral 50 mg daily dose, 3 capsules per dose during a six week treatment period.
  Arms: 50 mg
Drug: Placebo — oral placebo daily dose, 3 capsules per dose during a six week treatment period.
  Arms: Placebo

SUMMARY:
In a Phase II trial in subjects with nonrestorative sleep, PD 0200390 demonstrated a positive treatment effect relative to placebo on the primary endpoint, the weekly version of the Restorative Sleep Questionnaire (RSQ-W). In this study, the dose-response relationship of varying doses of PD 0200390 using the Restorative Sleep Questionnaire (RSQ-W), will be explored in Nonrestorative Sleep subjects.

ELIGIBILITY:
Inclusion Criteria:

* Awake unrestored or unrefreshed, associated with significant distress or impairment in social, occupational, or other important areas of functioning during the daytime, for at least 3 nights for the past 3 months prior to screening
* Self-report wake after sleep onset <45 mins for past 3 mos; self-report latency to sleep onset <20 mins for past 3 mos
* PSG (Polysomnography) sleep criteria of wake after sleep onset < 45 mins; Latency to persistent sleep <20 mins.

Exclusion Criteria:

* MAP (Multivariable Apnea Risk index) index > or = 0.5 at screening
* BMI = or > 32 kg/m2
* History or presence of breathing related disorders
* PSG findings consistent with and periodic limb movement disorder, narcolepsy or other dyssomnia or parasomnia including apnea-hypopnea index > 10/hr; or period limb movement with arousal index > 10/hr.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 306 (Actual)
Dates: Start 2008-04; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Total score of how an individual rates the restorative value of his/her sleep in the morning using the weekly version of the Restorative Sleep Questionnaire (RSQ-Weekly) | Weekly

SECONDARY OUTCOMES:
Measure sleep and early morning behavior during treatment using the Leeds Sleep Evaluation Questionnaire | Weeky
Total score of the Daily Restorative Sleep Questionnaire | Daily
Total score of the Multidimensional Assessment of Fatigue (MAF) | Weekly
Total score of the Sheehan Disability Scale to measure functional impairment | Weekly
Measure of health status using the Medical Outcomes Study Short Form-36 (SF-36v2-Acute) | Weekly
Total mood disturbance score using the Profile of Mood State-Short Form Questionnaire (POMS-SF) | Weekly
Total score of the Endicott Work Productivity Scale (EWPS) measuring work productivity. | Weekly
Disease severity and change using the Clinical Global Impression of Severity (CGI-S) as rated by the Clinician. | Weekly
Disease change (patient rated) measure using the Patient Global Impression of Change (PGIC). | Weekly

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (53):
- United States (48):
  - Pfizer Investigational Site, Glendale, Arizona
  - Pfizer Investigational Site, Phoenix, Arizona
  - Pfizer Investigational Site, Tucson, Arizona
  - Pfizer Investigational Site, Little Rock, Arkansas
  - Pfizer Investigational Site, Los Angeles, California
  - Pfizer Investigational Site, Pasadena, California
  - Pfizer Investigational Site, San Diego, California
  - Pfizer Investigational Site, San Francisco, California
  - Pfizer Investigational Site, Tustin, California
  - Pfizer Investigational Site, Wheat Ridge, Colorado
  - Pfizer Investigational Site, North Haven, Connecticut
  - Pfizer Investigational Site, Wallingford, Connecticut
  - Pfizer Investigational Site, DeLand, Florida
  - Pfizer Investigational Site, Miami, Florida
  - Pfizer Investigational Site, Naples, Florida
  - Pfizer Investigational Site, Orange City, Florida
  - Pfizer Investigational Site, Orlando, Florida
  - Pfizer Investigational Site, Pembroke Pines, Florida
  - Pfizer Investigational Site, South Miami, Florida
  - Pfizer Investigational Site, Atlanta, Georgia
  - Pfizer Investigational Site, Gainesville, Georgia
  - Pfizer Investigational Site, Chicago, Illinois
  - Pfizer Investigational Site, Indianapolis, Indiana
  - Pfizer Investigational Site, Overland Park, Kansas
  - Pfizer Investigational Site, Crestview Hills, Kentucky
  - Pfizer Investigational Site, Lexington, Kentucky
  - Pfizer Investigational Site, Baton Rouge, Louisiana
  - Pfizer Investigational Site, Chevy Chase, Maryland
  - Pfizer Investigational Site, Brighton, Massachusetts
  - Pfizer Investigational Site, North Dartmouth, Massachusetts
  - Pfizer Investigational Site, Chesterfield, Missouri
  - Pfizer Investigational Site, St Louis, Missouri
  - Pfizer Investigational Site, Las Vegas, Nevada
  - Pfizer Investigational Site, West Seneca, New York
  - Pfizer Investigational Site, Cary, North Carolina
  - Pfizer Investigational Site, Raleigh, North Carolina
  - Pfizer Investigational Site, Salisbury, North Carolina
  - Pfizer Investigational Site, Winston-Salem, North Carolina
  - Pfizer Investigational Site, Cincinnati, Ohio
  - Pfizer Investigational Site, Oklahoma City, Oklahoma
  - Pfizer Investigational Site, Clarks Summit, Pennsylvania
  - Pfizer Investigational Site, Uniontown, Pennsylvania
  - Pfizer Investigational Site, Warwick, Rhode Island
  - Pfizer Investigational Site, West Warwick, Rhode Island
  - Pfizer Investigational Site, Columbia, South Carolina
  - Pfizer Investigational Site, Austin, Texas
  - Pfizer Investigational Site, Dallas, Texas
  - Pfizer Investigational Site, Irving, Texas
- Canada (5):
  - Pfizer Investigational Site, Kelowna, British Columbia
  - Pfizer Investigational Site, Etobicoke, Ontario
  - Pfizer Investigational Site, Kitchener, Ontario
  - Pfizer Investigational Site, Parry Sound, Ontario
  - Pfizer Investigational Site, Toronto, Ontario

REFERENCES:
- [Derived] Drake CL, Hays RD, Morlock R, Wang F, Shikiar R, Frank L, Downey R, Roth T. Development and evaluation of a measure to assess restorative sleep. J Clin Sleep Med. 2014 Jul 15;10(7):733-41, 741A-741E. doi: 10.5664/jcsm.3860. PMID 25024650
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A4251033&StudyName=A%20Double-blind%2C%20Parallel%20group%2C%20Placebo-Controlled%20Outpatient%20Trial%20of%20PD%2000200390%20in%20Adults%20with%20Nonrestorative%20Sleep